CLINICAL TRIAL: NCT03481244
Title: Treatment of Adenovirus Disseminated Infections in Hematopoietic Stem Cell Transplant Patients With Adenovirus Digestive Replication- A Pharmaco-epidemiological Prospective Study
Brief Title: Treatment of Adenovirus Disseminated Infections in Hematopoietic Stem Cell Transplant Patients With Adenovirus Digestive Replication
Acronym: ADENOCLEAR
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: K140902J
Record Dates: First submitted 2018-03-22; First posted 2018-03-29 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Patients Who Underwent Allograft

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — stool specimens for ADN of adenovirus
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Disseminated Adv infections are associated with high morbidity and mortality in HSCT pediatric patients. The most common source of Adv infection after pediatric HSCT is the host digestive tract where latent Adv are reactivated after engraftment. We have shown in a monocentric study that Adv viral load in stools is a predictive factor of blood infection in children with digestive Adv infections. We assume that an early treatment, with antiviral drugs, such as cidofovir and brincidofovir, may avoid severe Adv infections and diseases and thus that molecular surveillance in stool is a critical factor for the control of Adv reactivations.

The study has two main objectives: (i) confirming the impact of Adv viral load in stools on the occurrence of blood infection based on a multicentric prospective cohort study design; and (ii) determining the prognostic and predictive factors for efficacy and toxicity of antiviral drugs, such as brincidofovir and cidofovir.

ELIGIBILITY:
Inclusion Criteria:

* Allogeneic hematopoietic stem cell transplantation from any donor other than full-matched related donor
* Age above 2 months and under 20 years
* Provide written informed consent from the parents (if <18) and child
* Free, informed and written consent, signed by the patient and investigator before any Study examination. If the patient is a minor by child (if possible) and both parents or child and the legal representative in case only one parent is alive

Exclusion Criteria:

* Hematopoietic stem cell transplantation from full-matched related donor
* Females who are pregnant or currently nursing
* Any patient receiving cidofovir, ribavirin or any other anti-viral drug under development given in order to treat or prevent
* Current disease attributed to adenovirus infection
* Lack of affiliation to a social security scheme (as a beneficiary or assignee).Current disease attributed to adenovirus infection

Ages: 2 Months to 20 Years | Sex: All
Age Groups: Child, Adult
Study Population: any patient age above 2 month- and under 20 year- old receiving an allogeneic hematopoietic stem cell transplant
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
rate of Adv blood infection according to levels of Adv DNA in stool samples. | 100 days
  Adv blood infection is defined as plasma Adv DNA level greater than 200 copies per milliliter
rate of response to antiviral drugs | 100 days
  Success will be defined as undetectable level of DNA of Adv in blood after a maximum of 4 weeks of treatment. After 4 weeks of treatment any detectable level of Adv DNA will be considered as a failure.

SECONDARY OUTCOMES:
Adv DNA levels > 5 log10 copies/ml in stool | 100 days
  measured at the end of treatment
Time required achieving 50% decrease of Adv load and undetectable Adv DNA. | 100 days
Time required achieving 90% decrease of Adv load and undetectable Adv DNA. | 100 days
Incidence of Adv probable or proven disease | 100 days
  We will use the definitions recommended by ECIL (detailed in Appendix 1).
  * Digestive infection: positive Adv PCR in stool
  * Local infection: positive Adv PCR in biopsy material or body fluids other than peripheral blood.
  * Systemic infection/viremia: positive Adv PCR in peripheral blood.
  * Probable disease: Adv infection plus corresponding symptoms and signs without histological confirmation.
  * Proven disease: Adv infection plus corresponding symptoms related to the infection and histological confirmation of Adv in the appropriate location.
Incidence of diarrhea | 100 days
Incidence of acute digestive graft versus host disease (aGvHD) | 100 days
Overall survival. | 100 days
Incidence of Adv probable or proven disease | 100 days
Genotypic analysis of the Adv DNA polymerase | 100 days
Detection and quantification of herpesviruses in blood | 100 days